CLINICAL TRIAL: NCT00239382
Title: A Randomized, Open-labelled Study to Compare the Efficacy and Safety of Meloxicam 15 mg IM Ampoules Once Daily and Meloxicam 15 mg Tablets Administered Orally Once Daily Over a Period of 7 Days in Patients With RA.
Brief Title: A Study to Compare Meloxicam IM Once Daily Versus Meloxicam Orally Once Daily in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 107.266
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Meloxicam

INTERVENTIONS:
Drug: Meloxicam ampoule
Drug: Meloxicam tablet

SUMMARY:
The objective of this trial was to assess the efficacy and safety of 15 mg meloxicam i.m. once daily compared with 15 mg meloxicam tablets once daily p.o. in patients with Rheumatoid arthritis over a time period of 7 days.

DETAILED DESCRIPTION:
This was a randomized (1:1), open-label, multi-center, active-control, parallel-group study to compare the efficacy of 15 mg meloxicam i.m. once daily compared with 15 mg meloxicam tablets once daily p.o. in patients with rheumatoid arthritis over a time period of 7 days.

Patients eligible for the trial who met all inclusion and exclusion criteria and who gave their informed consent were randomized to one of two treatment groups (i.e. meloxicam ampoule or meloxicam tablet).

The study period totaled 8-14 days included screening, randomisation, study drug administration, and 7-day follow-up. The relevant assessment were performed on the day of randomisation and 7-day follow up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or above
* The patient has rheumatoid arthritis, as defined by the American Rheumatism Association.
* Assessment of overall pain (by the patient), after a washout for NSAID of at least 2 days (3 days for oxicams), must exceed 40 mm on a 100 mm visual analogue scale (VAS)
* Symptoms of RA requiring administration of NSAIDs
* Outpatients
* Willingness and ability to provide written informed consent.

Exclusion Criteria:

* Known or suspected hypersensitivity to the trial drugs or their excipients, analgesics, antipyretics or NSAIDs
* Any clinical evidence of active peptic ulceration during the previous 6 months
* Pregnancy or breastfeeding (precaution: attention should be drawn to reports that NSAIDs were reported to decrease the effectivity of intrauterine devices)
* Asthma, nasal polyps, angioneurotic oedema or urticaria following the administration of aspirin or NSAIDs
* Concomitant treatment with anti-coagulants (including heparin), lithium
* Concomitant administration of other NSAIDs or analgesic agents (except paracetamol up to 4g/day)
* Administration of any NSAID during the last 2 days (3 days for any oxicam) prior to the first administration of the trial drug
* Concomitant treatment with methotrexate, sulfasalazine, D-penicillamine, chloroquine or any other disease modifying antirheumatic drug initiated or with an altered dose over the previous 3 months
* Concomitant treatment with an oral corticosteroid initiated or with an altered dose over the previous month
* Parenteral or intraarticular administration of corticosteroids in the previous month
* Any i.m. injection during the previous 7 days
* Synovectomy and/or surgical treatment for RA in the previous month or during the trial
* Any physiotherapy which will be changed during the trial
* Any contra-indication to i.m. injections
* Clinical evidence of or known severe cardiac, hepatic, renal, metabolic, haematological disease, mental disturbance, ulcerative colitis
* Any other rheumatological or non-rheumatological disease that could interfere with the evaluation of efficacy and safety
* Serum creatinine 125 % of the upper limit of normal range ; aspartate amino-transferase (AST/SGOT) and/or alaline amino-transferase (ALT/SGPT) 200 % of the upper limit of normal range
* Platelet count < 100,000/mm3 ; leucocytes count < 3,000/mm3
* Participation in another clinical trial during this study or during the previous month
* Previous participation in this trial (i.e. having been allocated a randomized treatment number)
* Patient unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-07-01 (Actual); Primary Completion 2004-12-01 (Actual); Study Completion 2004-12-31 (Actual)

PRIMARY OUTCOMES:
Patient's assessment of overall pain | 7 days
Patient's global assessment of disease activity | 7 days

SECONDARY OUTCOMES:
Investigator's Global Assessment of Disease Activity | 7 days
Tender/Painful Joint Count | 7 days
Swollen Joint Count | 7 days
Duration of Morning Stiffness | 7 days
Patient's assessment of physical function | 7 days
Final Global Assessment of Efficacy by Patient | 7 days
Final Global Assessment of Efficacy by Investigator | 7 days
Withdrawals due to Inadequate Efficacy | 7 days
Change in Patient Status With Regard to Arthritic Condition as Assessed by the Patient | 7 days
Change in Patient Status With Regard to Arthritic Condition as Assessed by the Investigator | 7 days
Onset of Analgesic Action | 7 days
Time to Maximum Pain Relief After the First Trial Drug Administration | 7 days
Paracetamol Consumption | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Shanghai
Locations (8):
- China (8):
  - People's Hospital, Beijing University, Beijing
  - Beijing Xuan Wu Hospital, Beijing
  - 1st Affiliated, Anhui Medical University, Hefei City, Anhui Province
  - Qilu Hospital, Shang Dong University, Nanzhou
  - Shanghai Renji Hospital, Shanghai
  - Shanghai Zhongshan Hospital, Shanghai
  - Shanghai Guanghai Hospital, Shanghai
  - Shanghai Changhai Hospital, Shanghai